CLINICAL TRIAL: NCT02346643
Title: BINGO: A Post Market Evaluation of Chronic intractaBle paIN and the Efficacy of drG stimulatiOn in the Nordic Region
Brief Title: A Post Market Evaluation of Chronic intractaBle paIN and the Efficacy of drG stimulatiOn in the Nordic Region
Acronym: BINGO
Status: Terminated | Type: Observational
Why Stopped: Budget Allocation Decision by Sponsor
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-SMI-2013
Record Dates: First submitted 2015-01-07; First posted 2015-01-27 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated Subjects: All subjects recruited and treated with the Axium neurostimulator
  Interventions: Device: Implantation with the commercially available Axium Neurostimulator

INTERVENTIONS:
Device: Implantation with the commercially available Axium Neurostimulator

SUMMARY:
11-SMI-2013 is a post market, observational, questionnaire based study to assess the effectiveness of the commercially available Axium neurostimulator in the management of intractable, chronic pain

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Chronic, intractable pain for at least 6 months
4. Failed conservative treatments for chronic pain including but not limited to pharmacological therapy, physical therapy and interventional pain procedures for chronic pain
5. Minimum baseline pain rating of 60 mm on the VAS in the primary region of pain
6. Subject is able to provide written informed consent

Exclusion Criteria:

1. Female subject of childbearing potential is pregnant/nursing or plans to become pregnant during the study duration
2. Escalating or changing pain condition within the past month as evidenced by investigator examination
3. Subject has had corticosteroid therapy at an intended site of stimulation within the past 30 days
4. Subject has had radiofrequency treatment of an intended target DRG within the past 3 months
5. Subject currently has an active implantable device including ICD, pacemaker, spinal cord stimulator or intrathecal drug pump
6. Subject is unable to operate the device
7. Subjects currently has an active infection
8. Subject has participated in another clinical investigation within 30 days
9. Subject has a coagulation disorder or uses anticoagulants that, in the opinion of the investigator, precludes participation
10. Subject has been diagnosed with cancer in the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Pain Patients
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Akademiska sjukhuest, Uppsala

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Subjects: All subjects enrolled into the study with intent to treat with the Axium Neurostimulator
Period: Overall Study
Arm/Group | All Enrolled Subjects
Started | 41
Received Trial System | 29
Received Permanent System (Two cases were trials on the table (all-in-one procedures)) | 31
Completed | 6
Not Completed | 35

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 41
Age, Continuous [Mean (Full Range); unit: years] | 47 [20 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 41

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity in Primary Region of Pain
Description: Assessed by Change in Pain Intensity on a Visual Analogue Scale (VAS) from Pre-Treatment Baseline.
  The Visual Analog Scale (VAS) is self-administered instrument assessing average pain intensity. Subjects rated their pain on a horizontal line, 10 cm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher pain level. The values range from 0 (minimum pain) to 10 (maximum pain).
Time Frame: Post treatment at 3, 6 and 12 months
Population: Differences in participants over time is due to early withdrawals and missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Subjected Treated With the Permanent: All subjects treated with the Axium implantable neurostimulator
Arm/Group | Subjected Treated With the Permanent
Number analyzed (Participants) | 31
units on a scale
  Baseline | 7.6 (1.3)
  3-Month Visit: number analyzed (Participants) | 27
  3-Month Visit | 4.9 (2.4)
  6-Month Visit: number analyzed (Participants) | 25
  6-Month Visit | 5.3 (2.7)
  12-Month Visit: number analyzed (Participants) | 18
  12-Month Visit | 4.8 (2.8)

2. Primary Outcome: Pain Intensity in Overall Pain
Description: Assessed by Change in Pain Intensity on a Visual Analogue Scale (VAS) from Pre-Treatment Baseline
  The Visual Analog Scale (VAS) is self-administered instrument assessing average pain intensity. Subjects rated their pain on a horizontal line, 10 cm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher pain level. The values range from 0 (minimum pain) to 10 (maximum pain).
Time Frame: Post treatment at 3, 6 and 12 months
Population: Differences in participants over time is due to early withdrawals and missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjected Treated With the Permanent
Number analyzed (Participants) | 31
units on a scale
  Baseline | 7.5 (1.5)
  3-Month Visit: number analyzed (Participants) | 27
  3-Month Visit | 5.3 (2.3)
  6-Month Visit: number analyzed (Participants) | 25
  6-Month Visit | 5.4 (2.8)
  12-Month Visit: number analyzed (Participants) | 18
  12-Month Visit | 5.6 (2.3)

ADVERSE EVENTS:
Arm/Group | All Enrolled Subjects
Serious Adverse Events (participants affected / at risk) | 1/41
Other Adverse Events (participants affected / at risk) | 7/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=41)
Post-dural puncture headache (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=41)
IPG Pocket Pain (Injury, poisoning and procedural complications) | 1 (1)
High Lead Impedance (Investigations) | 1 (1)
Loss of Stimulation (Injury, poisoning and procedural complications) | 2 (2)
Lead Severed (Injury, poisoning and procedural complications) | 1 (1)
Pain at Incision Site (Injury, poisoning and procedural complications) | 2 (2)
Arrhythmia and Irregularities (Cardiac disorders) | 1 (1)
Back Pain (General disorders) | 1 (1)
Erythema or Drainage or Inflammation (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Gluteal muscle pain (Injury, poisoning and procedural complications) | 1 (1)
Upper Extremities Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days